CLINICAL TRIAL: NCT04209127
Title: Single Blinded Randomized Controlled Study of Symptom Improvement After Uterine Artery Embolization (UAE) Versus Ultrasound Guided Percutaneous/transvaginal Microwave Ablation, Evaluated by Validated Questionnaires
Brief Title: Comparing Efficacy of Microwave Vs Embolization Treatment for Adenomyosis
Acronym: ADENOMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, Senior Consultant, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADENOMIC1
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Uterine Artery Embolization; Ethanol

STUDY DESIGN:
Intervention Model Description: RCT with inteventional cohort continuation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microwave treatment (Experimental): Percutaneous or vaginal application of microwave antenna with microwave treatment for adenomyosis
  Interventions: Procedure: Microwave treatment via needle antenna
- Control (Active Comparator): Uterine artery embolization; percutaneous application of a catheter into the femoral artery or branches thereof
  Interventions: Procedure: Embolization of uterine artery or branches thereof (routine treatment where polyvinyl alcohol particles are released into the predefined bloodstream)

INTERVENTIONS:
Procedure: Microwave treatment via needle antenna — Microwave treatment via needle antenna, (Emprint Covidien microwave ablation system) either percutaneous or vaginally administrated
  Arms: Microwave treatment
Procedure: Embolization of uterine artery or branches thereof (routine treatment where polyvinyl alcohol particles are released into the predefined bloodstream) — Embolization via percutaneous catheter
  Arms: Control

SUMMARY:
Single blinded randomized controlled study of symptom improvement after uterine artery embolization (UAE) versus ultrasound guided percutaneous/transvaginal microwave ablation, evaluated by validated questionnaires.

Adenomyosis is a benign condition causing pain and bleeding disorders in many women. Hysterectomy has historically been the golden standard for treatment as well as (postoperatively) diagnosis of the disease. In accordance with refined diagnostic tools such as ultrasound and/or MRI, minimally invasive treatments for adenomyosis are being explored.

We plan to compare two minimally invasive techniques: embolization of the uterine artery (a commonly used procedure) and microwave ablation of adenomyotic tissue (previously only in clinical use in China).

DETAILED DESCRIPTION:
Single blinded randomized controlled study of symptom improvement after uterine artery embolization (UAE) versus ultrasound guided percutaneous/transvaginal microwave ablation, evaluated by validated questionnaires.

Background

Adenomyosis is a benign gynecological condition, where endometrial glands and stroma invades the myometrial walls of the uterus. The disease is thought to be estrogen-dependent, but the etiology, as well as the prevalence, is currently unknown. Known risk-factors are previous uterine surgery and parity, although the disease has been found also in nulligravida with no previous uterine trauma. Adenomyosis can cause severe dysmenorrhea, menorrhagia, chronic pelvic pain and infertility. Historically diagnosis has been made post hysterectomy by pathologists, however with transvaginal ultrasound (TVUS) as well as MRI the condition is now possible to identify with non-invasive methods.

Hysterectomy has previously been seen as the golden standard treatment for adenomyosis, but may cause long-term side effects such as genitovaginal prolapse. It also carries a substantial risk of short term complications such as infections and organ damage.

Symptomatic treatment such as the levonogestrel intrauterine system (LNG-IUS) can be effective, however there is a risk of expulsion and irregular bleedings.

In recent years, increasing attention has been paid to the study of minimally invasive or non-invasive therapies with uterine preservation such as uterine arterial embolization (UAE), radiofrequency (RF), microwave treatment and high intensity focused ultrasound (HIFU). A randomized controlled study is ongoing, comparing UAE and hysterectomy. RF ablation often requires the aid of a laparoscopic procedure, which is invasive. HIFU is currently only described in small cohorts and case-reports. Ultrasound or computer tomography guided percutaneous microwave thermal ablation is minimally invasive, has low time requirements, is easy to perform, and has been broadly used for the treatment of solid tumours in organs other than the uterus with favourable effects.

Microwave ablation of adenomyosis has been performed in China. The effect and acceptability has been high. The research team in this study has been to China to study the treatment. We have visited the clinic and studied the procedure as well as talked to patients pre- and post operatively . The equipment at Danderyd Hospital has the same output effects as the equipment in China. Danderyd Hospital has approved the method for use in uterine myomas. However, no randomized comparative study of other minimally invasive methods has been performed.

This study aims to compare the effectiveness, feasibility and acceptability of percutaneous CT- or ultrasound guided microwave ablation and uterine artery embolization for the treatment of adenomyosis in a randomized single blind study.

Recruitment and Randomization

Women fulfilling inclusion criteria and without exclusion criteria will be identified at the outpatient clinic of Danderyd Hospital. Advertisement may be placed in local newspapers or on social media (Facebook and Instagram) and relevant webpages or in gynecological clinics.

Women will be randomized after having been informed orally and in written and after having signed informed consent and after fulfilling inclusion and exclusion criteria after MRI-examination. Randomization will be in random permuted blocks of 6 at a ratio of 1:1. The randomization will be according to a computer generated randomization sequence. After patients have signed informed consent and fulfill inclusion without exclusion criteria after the initial magnetic resonance imaging they will be allocated to an intervention by consecutive opening of sealed opaque envelopes containing the randomization code.

Blinding

Patients and investigators will not be blinded. The MRI will be performed and evaluated by a blinded radiologist.

Method

Pre randomization evaluation After having signed informed consent but before randomization patients will undergo MRI of the uterus. Patients with endometriosis or a clinically significant presence of uterine fibroids (myomas>3cm) will be excluded.

All women included in the study after MRI examination will fill in a PBAC evaluation during the menses preceding treatment. Women will fill a VNRS for maximal pain during 1 month prior to treatment. In addition a full blood panel will be evaluated.

As for uterine artery embolization no pathologist report will be performed before any treatment.

Microwave ablation Microwave ablation will be performed percutaneously or vaginally using a Covidien Emprint microwave ablation system with a 30-80 Watts effect in 14-16 gauge needle with a ceramic tip using computer tomography with fusion technique or ultrasound for adenomyosis imaging and needle guidance. After identification of the needle path with CT or peroperative ultrasound a small skin incision using a scalpel will made for the needle entry in the case of percutaneous treatment. No incision will be made if treatment is given vaginally. When needed to optimize the needle path in order not to damage adjacent organs, artificial ascites (approx 500mL Ringer-acetate) will be created using a thin syringe through the abdominal wall. The ablation zone of a 70W needle is estimated to be 4x3x3 cm after 300s or 5x4x4 cm after 600s. Patients will be given intravenous anesthesia with spontaneous breathing or general anesthesia during treatment to minimize movement during ablation.

Uterine artery embolization Embolization will be performed in conscious women with an epidural catheter or patient controlled analgesia for pain relief. A catheter will be inserted in the femoral artery to access the uterine artery during x-ray monitoring and during administration of contrast to visualize the adenomyotic tissue and its supporting arterial supply. When the supporting arterial branch has been identified polyvinyl alcohol particles are released into the bloodstream. These particles cause a thrombosis in the vessel.

Evaluation post treatment Women will estimate VNRS maximum postoperative pain day of surgery and the following 7 days. In addition, they will note how many days passed before all pain subsided, use of pain medication will be noted and period until resuming normal daily activities. The period of hospitalization will be noted.

Menstrual blood loss (PBAC) will be noted the first menstruation, menstruation number 3 and 5 post treatment. PBAC is a validated instrument for menstrual blood loss quantification. UFS-QOL is a validated instrument for women with uterine fibroids, but is commonly used also in trials regarding adenomyosis, and will be evaluated 6 months post treatment.

Follow-up visits will be after 1-2 menstruation at approximately 2 months and at 6 months post-treatment.

At follow up visit 2 months (+/-2 weeks) and 6 months (+/-2 weeks) post treatment acceptability will be assessed as overall satisfaction of treatment on a scale from 1-7 and if the woman would recommend the treatment to a friend. At the follow up visit at 6 months hemoglobin, cancer antigen 125 (CA-125), Anti-Müllerian Hormone (AMH), and prolactine (PRL) will be measured. AMH estimates the effect of the treatment on the ovarian reserve. CA-125 and PRL have been used to evaluate pathophysiological changes in adenomyosis. These will be compared to levels taken on the day of the operative procedure. A uterine biopsy will also be performed.

A new MRI scan will be performed 6 months post treatment (+/-21 days). Women will then be asked to participate in a long-term follow up (>12 months) with evaluation of recurrence of symptoms, with clinical controls (gynecological exams and TVUS) and using PBAC and UFS-QOL yearly until retraction of consent.

Continuation of the study:

During our analysis of the initial pilot study, we noticed significant alleviation of symptoms in both treatment groups, however no significant difference between the groups (MWA vs UAE).

We however noted a significant better postoperative outcome in the MWA group:

hospitalization, return to ADL and need of analgesics postoperatively were all strongly in favor of MWA.

Also, the international research on MWA and fertility wish has proceeded during our initial study period, suggesting no significant higher risk for adverse oucomes in pregnancies after MWA.

These altered conditions made us apply for a continuation of the study to the Regional Ethical Review Board of Stockholm, with the following design:

* Prospective Interventional study of MWA treatment for symptomatic adenomyosis, n=50
* All patients receive MWA treatment and follow-up after 6 months
* Inclusion criterias remain unchanged, except for MRI no longer needed for diagnostics
* Fertility wish, cocurrent myomas and/or endometriosis no longer an exlusion criteria

Primary and secondary outcomes remain unchanged. Due to reasons listed above, we have now expanded the study period until June 2026.

Clinical significance

Adenomyosis is a benign condition but have a significant impact on the lives of women, and the condition is not well studied. Reports have suggested adenomyosis in approximately 40% of patients undergoing hysterectomy. Women with adenomyosis are much more likely to report on symptoms as dysmenhorrea, heavy menstrual bleeding, infertility and chronic pelvic pain. As hysterectomy is a highly invasive procedure with costs for women in terms of absence from work and short and long term complications, finding new minimally invasive and uterine-sparing treatments would be beneficial for affected women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 30-55 with symptomatic adenomyosis
* Premenopausal
* Adenomyosis diagnosted by TVUS
* Willing to comply with protocol

Exclusion Criteria:

* Body Mass Index >35
* Treatment with anticoagulant/bleeding disorder
* Contraindication for UAE or general anesthesia

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
1. Symptom improvement 6 months post treatment (+/-21 days) compared to pre treatment, evaluated by UFS-QOL - The score on Symptom Severity Scale | 6 months
  Symptom improvement evaluated by the validated questionnaire UFS-QOL, which is subdivided into Symptom Severity Scale (0-100, where higher number represent worsened symptoms) and HRQL items (concern, activities, energy/mood, control, self-consciousness and sexual function, range 0-100 where higher numbers represent better Quality of Life)

SECONDARY OUTCOMES:
Reduction of adenomyosis by imaging | 6 months
  Reduction of uterus volume/adenomyosis affected areas, measured as lesional size (in mm or cm) measured by Transvaginal ultrasound and/or MRI
Hospitalization | Up to 8 weeks post treatment
  How long time (in days) the patient needed postoperative care in the ward, identified by the patients Medical chart
Sick leave | Up to 8 weeks post treatment
  How many Days until the patient resumed normal working hours
Pain medication | Up to 8 weeks post treatment
  How much and what type of pain medication the patient needed post operatively
Acceptability | 2 months and 6 months post treatment
  Patients description wether they would recommend the treatment to a friend, measured by a 7-point Likert scale (1-7, where higher number represents a greater acceptability)
Symptom improvement 6 months post treatment (+/-21 days) compared to pre treatment, evaluated by PBAC (pictorial blood loss assessment chart) | 6 months
  Symptom improvement in regard to menstrual blood loss, PBAC ranges from 0->4000 and cut-off for the diagnose of Heavy Menstrual Bleeding is normally PBAC>100
Symptom improvement 6 months post treatment (+/-21 days) compared to pre treatment, evaluated by | 6 months
  Symptom improvement in regard to menstrual pain, evaluated by VNRS (0-10, recorded each day of the menstrual period, where 0 is no pain and 10 worst possible pain)
1. Symptom improvement 6 months post treatment (+/-21 days) compared to pre treatment, evaluated by UFS-QOL - The Health related quality of life score | 6 months
  Symptom improvement evaluated by the validated questionnaire UFS-QOL, which is subdivided into Symptom Severity Scale (0-100, where higher number represent worsened symptoms) and HRQL items (concern, activities, energy/mood, control, self-consciousness and sexual function, range 0-100 where higher numbers represent better Quality of Life)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kopp Kallner, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Struble J, Reid S, Bedaiwy MA. Adenomyosis: A Clinical Review of a Challenging Gynecologic Condition. J Minim Invasive Gynecol. 2016 Feb 1;23(2):164-85. doi: 10.1016/j.jmig.2015.09.018. Epub 2015 Sep 30. PMID 26427702
- [Background] Pinzauti S, Lazzeri L, Tosti C, Centini G, Orlandini C, Luisi S, Zupi E, Exacoustos C, Petraglia F. Transvaginal sonographic features of diffuse adenomyosis in 18-30-year-old nulligravid women without endometriosis: association with symptoms. Ultrasound Obstet Gynecol. 2015 Dec;46(6):730-6. doi: 10.1002/uog.14834. PMID 25728241
- [Background] Dueholm M. Uterine adenomyosis and infertility, review of reproductive outcome after in vitro fertilization and surgery. Acta Obstet Gynecol Scand. 2017 Jun;96(6):715-726. doi: 10.1111/aogs.13158. PMID 28556124
- [Background] Li X, Liu X, Guo SW. Clinical profiles of 710 premenopausal women with adenomyosis who underwent hysterectomy. J Obstet Gynaecol Res. 2014 Feb;40(2):485-94. doi: 10.1111/jog.12211. Epub 2013 Oct 22. PMID 24148010
- [Background] Van den Bosch T, Van Schoubroeck D. Ultrasound diagnosis of endometriosis and adenomyosis: State of the art. Best Pract Res Clin Obstet Gynaecol. 2018 Aug;51:16-24. doi: 10.1016/j.bpobgyn.2018.01.013. Epub 2018 Feb 14. PMID 29506961
- [Background] Sheng J, Zhang WY, Zhang JP, Lu D. The LNG-IUS study on adenomyosis: a 3-year follow-up study on the efficacy and side effects of the use of levonorgestrel intrauterine system for the treatment of dysmenorrhea associated with adenomyosis. Contraception. 2009 Mar;79(3):189-93. doi: 10.1016/j.contraception.2008.11.004. Epub 2008 Dec 11. PMID 19185671
- [Background] de Bruijn AM, Smink M, Lohle PNM, Huirne JAF, Twisk JWR, Wong C, Schoonmade L, Hehenkamp WJK. Uterine Artery Embolization for the Treatment of Adenomyosis: A Systematic Review and Meta-Analysis. J Vasc Interv Radiol. 2017 Dec;28(12):1629-1642.e1. doi: 10.1016/j.jvir.2017.07.034. Epub 2017 Oct 9. PMID 29032946
- [Background] de Bruijn AM, Lohle PN, Huirne JA, de Vries J, Twisk M; QUESTA-Trial Group; Hehenkamp WJ. Uterine Artery Embolization Versus Hysterectomy in the Treatment of Symptomatic Adenomyosis: Protocol for the Randomized QUESTA Trial. JMIR Res Protoc. 2018 Mar 1;7(3):e47. doi: 10.2196/resprot.8512. PMID 29496654
- [Background] Guo Q, Xu F, Ding Z, Li P, Wang X, Gao B. High intensity focused ultrasound treatment of adenomyosis: a comparative study. Int J Hyperthermia. 2018;35(1):505-509. doi: 10.1080/02656736.2018.1509238. Epub 2018 Oct 11. PMID 30306813
- [Background] Hai N, Zhang J, Xu R, Han ZY, Liu FY. Percutaneous microwave ablation with artificial ascites for symptomatic uterine adenomyosis: initial experience. Int J Hyperthermia. 2017 Sep;33(6):646-652. doi: 10.1080/02656736.2017.1285444. Epub 2017 Feb 15. PMID 28118773
- [Background] Xu RF, Zhang J, Han ZY, Zhang BS, Liu H, Li XM, Ge HL, Dong XJ. Variables associated with vaginal discharge after ultrasound-guided percutaneous microwave ablation for adenomyosis. Int J Hyperthermia. 2016 Aug;32(5):504-10. doi: 10.3109/02656736.2016.1150523. Epub 2016 Apr 18. PMID 27087631
- [Background] Yang Y, Zhang J, Han ZY, Ma X, Hao YL, Xu CT, Xu RF, Zhang BS. Ultrasound-guided percutaneous microwave ablation for adenomyosis: efficacy of treatment and effect on ovarian function. Sci Rep. 2015 May 5;5:10034. doi: 10.1038/srep10034. PMID 25942631
- [Background] Xia M, Jing Z, Zhi-Yu H, Jian-Ming C, Hong-Yu Z, Rui-Fang X, Yu Y, Yan-Li H, Bao-Wei D. Feasibility study on energy prediction of microwave ablation upon uterine adenomyosis and leiomyomas by MRI. Br J Radiol. 2014 Aug;87(1040):20130770. doi: 10.1259/bjr.20130770. Epub 2014 Jun 20. PMID 24947033
- [Background] Zhang J, Han ZY, Feng L, Wang F, Hu DM, Wen B, Li ZC. [Ultrasound-guided percutaneous microwave ablation in the treatment of diffuse adenomyosis]. Zhonghua Yi Xue Za Zhi. 2011 Oct 25;91(39):2749-52. Chinese. PMID 22322052
- [Background] Reid PC, Coker A, Coltart R. Assessment of menstrual blood loss using a pictorial chart: a validation study. BJOG. 2000 Mar;107(3):320-2. doi: 10.1111/j.1471-0528.2000.tb13225.x. PMID 10740326
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Harding G, Coyne KS, Thompson CL, Spies JB. The responsiveness of the uterine fibroid symptom and health-related quality of life questionnaire (UFS-QOL). Health Qual Life Outcomes. 2008 Nov 12;6:99. doi: 10.1186/1477-7525-6-99. PMID 19014505
- [Background] Coyne KS, Margolis MK, Murphy J, Spies J. Validation of the UFS-QOL-hysterectomy questionnaire: modifying an existing measure for comparative effectiveness research. Value Health. 2012 Jul-Aug;15(5):674-9. doi: 10.1016/j.jval.2012.03.1387. Epub 2012 Jun 8. PMID 22867776